CLINICAL TRIAL: NCT03193216
Title: The Impact of Adjuvant Liquid Alginate on Endoscopic Ablation Therapy of Complicated Barrett's Esophagus: A Pilot Study
Brief Title: The Impact of Adjuvant Liquid Alginate on Endoscopic Ablation Therapy of Complicated Barrett's Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00065861
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Barretts Esophagus With Dysplasia
Keywords: Barrett's; GERD; reflux; alginate solution; proton pump inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Alginates

STUDY DESIGN:
Intervention Model Description: This is a pilot prospective cohort study at a single tertiary center who will be compared to historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alginate group (Experimental): Patients in this group will be taking the study medication -- alginate solution in addition to standard of care twice daily proton pump inhibitor therapy
  Interventions: Drug: Alginates

INTERVENTIONS:
Drug: Alginates — Liquid Alginate therapy will be added to twice daily PPI regimen. Patients will be asked to take the alginate solution four times daily (following meals and at bedtime) at 10ml/dose.
  Other Names: Gaviscon Advance

SUMMARY:
This study evaluates the addition of an alginate based solution to twice daily proton pump inhibitor therapy (PPI) in patients undergoing ablative therapy for dysplastic Barrett's esophagus. The investigators hypothesize that the addition of this medication will help to achieve complete remission of Barrett's over a shorter period of time.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a pre-cancerous condition in the esophagus that results from constant acid exposure and is a precursor to esophageal adenocarcinoma (EAC). Surprisingly, EAC rates continue to rise despite efforts aimed at addressing BE. Patients with dysplastic BE are at increased risk for developing EAC and in high grade dysplasia (HGD), this risk can be as high as 6% per year. For these reasons, these patients are candidates for ablation therapy, either with cryotherapy, endoscopic mucosal resection (EMR), and/or radiofrequency ablation (RFA). In patients receiving ablative therapy, 3-5 treatments are typically required before there is resolution of all Barrett's epithelium while patients remain on twice daily proton pump therapy.

A recent case study by the current authors demonstrated initial failed response of BE with HGD to RFA and subsequently cryotherapy. Only after initiation of a liquid alginate solution (Gaviscon Advance - UK formulation) was there a subsequent rapid and complete response to therapy. This case suggests that liquid alginate provided additional esophageal protection allowing mucosal healing and an overall enhanced response to treatment. This finding is mechanistically plausible given existing evidence demonstrating the carcinogenic properties of bile acids and injurious activity of pepsin in non-acid refluxate, and liquid alginate's unique ability to control these components and inhibit acid reflux. The investigators feel further investigation is warranted in studying the role of adjunct liquid alginate solution in patients undergoing treatment for BE.

The ingredient of interest in is alginic acid (alginate), a polysaccharide found in the cell walls of brown algae. Alginates are unique in their ability to form a protective layer above gastric contents upon exposure to gastric acid, thus limiting exposure of esophageal epithelium to gastric acid, bile acid, pepsin, and other parts of the gastric contents. Concurrently, the bicarbonate in alginate-based solutions forms carbon dioxide in the presence of gastric acid, which converts the gel into foam which floats to the surface of the gastric contents. Hence, alginate solutions form "rafts" which provide a physical barrier to acid reflux, as well as a pH-neutral substitute which refluxes preferentially over gastric acid.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18 (2) Biopsy-proven complicated BE (low/high grade grade dysplasia or IMC, confirmed by our institution's GI pathologist) As part of standard of care, all patients' biopsies will be confirmed with the institutions' GI pathologist and, either with outside biopsies or from biopsies completed at the primary institution.

Exclusion Criteria:

* 1) Moderate to severe renal impairment, as defined by eGFR< 60 for 2 consecutive readings (2) Lack of capacity for decision-making (3) Allergy to hydroxybenzoates (4) Patients with uncontrolled hypertension or decompensated heart failure (5) Pregnancy- patients of child-bearing potential will be tested. (6) Patients with elevated calcium or potassium on screening laboratory testing (labs completed within the last month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had two groups. An active group with participants receiving alginate along with EET treatment and a historical control group comprised of a historical cohort of patients with dysplastic Barrett's esophagus who had EET treatment from 2017 to 2020. All patients in the historical group were treated by the same expert endoscopists included in the study and were on twice a day PPI therapy alone. Patients were matched by age, race, and length of BE.
Groups:
- Historical Control Group: A control group comprised of a historical cohort of patients with dysplastic Barrett's esophagus undergoing EET treatment from 2017 to 2020 were collected.
Period: Overall Study
Arm/Group | Alginate Group | Historical Control Group
Started | 24 | 21
Completed | 14 | 21
Not Completed | 10 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Physician Decision | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alginate Group | Historical Control Group | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Full Range); unit: years] | 61.1 [27 to 74] | 64.9 [46 to 79] | 63 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 21 | 16 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 21 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 22 | 21 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Successful Eradication
Description: To compare the percentage of patients who achieved complete endoscopic eradication of dysplastic Barrett's Esophagus(BE) and non-dysplastic BE with the combination of PPI and liquid alginate solution vs. those treated with PPI alone within eighteen months from the start of treatment.
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Alginate Group | Historical Control Group
Number analyzed (Participants) | 14 | 21
percentage of participants
  Percentage of patients with eradication of dysplasia | 45.5 | 38.1
  Percentage of patients with eradication of all Barretts (dysplasic and non-dysplastic) | 36.4 | 19.04

2. Secondary Outcome: Number of Treatments (Mean)
Description: To compare the number of treatment sessions required to achieve endoscopic eradication of dysplastic BE and complete eradication of all BE (dysplastic and non-dysplastic) in patients treated with the combination of PPI and liquid alginate solution vs. those treated with PPI alone.The minimum number of treatments would be 1 and maximum number of treatments in the 18 month period is 8.
Time Frame: 18 months
Measure: Mean (Full Range); unit: number of treatment sessions
Arm/Group | Alginate Group | Historical Control Group
Number analyzed (Participants) | 14 | 21
number of treatment sessions
  Average number of treatments to achieve eradication of dysplasia | 3.1 [1 to 8] | 3.88 [1 to 8]
  Average number of treatments to achieve eradication of all Barrett's (dysplastic and non-dysplastic) | 3.75 [1 to 8] | 5 [1 to 8]

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected for eighteen months on each patient who was enrolled in the study. AE data was not collected for the historical control group since they were not actively enrolled onto the study, but their data from previous treatment was used to compare with the active participants.
Description: Definition does not differ.
Arm/Group | Alginate Group | Historical Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/0
Other Adverse Events (participants affected / at risk) | 0/22 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT03193216/Prot_SAP_000.pdf